CLINICAL TRIAL: NCT04756999
Title: The Effect of Foot Reflexology Applied to Dialysis Patients on Quality of Life and Symptom Control: A Randomized Clinical Trial
Brief Title: The Effect of Foot Reflexology Applied on Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gizem Göktuna, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Issue: 2020/29-48
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Nursing Caries
Keywords: reflexology; dialysis; nursing care
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant
Masking Description: Single Blind Randomised Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): informed consent forms, nine sessions of foot reflexology massage will be given to reflex points including the solar plexus, brain, pituitary, thyroid, diaphragm, upper lymphs, lung, spinal cord and adrenal glands for 3 weeks. Then data collection tools were applied.
  Interventions: Behavioral: massage therapy
- Control (Placebo Comparator): informed consent forms, foot massage were performed. Then data collection tools were applied.
  Interventions: Behavioral: massage therapy

INTERVENTIONS:
Behavioral: massage therapy — Reflexology is massage therapy used to maintain and improve health, as well as relieve some symptoms.

SUMMARY:
Reflexology is massage therapy used to maintain and improve health, as well as relieve some symptoms. Foot reflexology, which is thought to have an effect on dialysis symptoms, will be applied to hemodialysis patients in 9 sessions. In this study, it is aimed to determine the effect of foot reflexology applied to dialysis patients on sleep, anxiety and quality of life.

DETAILED DESCRIPTION:
Reflexology is defined as a holistic treatment based on stimulating the nerves and blood circulation in the body by manually stimulating the reflex points in the hands and feet corresponding to all parts of the body, organs and systems. In the literature, there are many studies conducted in different samples to evaluate the effectiveness of reflexology massage. Hemodialysis patients are also included in these samples. Hemodialysis patients are faced with many physical and emotional symptoms such as lifestyle changes, psychosocial effects, side effects due to treatment, during their treatment process. Nurses play an important role in alleviating and eliminating these complaints. Objective: It is aimed to determine the effect of foot reflexology applied to dialysis patients on sleep, anxiety and quality of life. Design: Randomized, controlled, prospective study. Setting: University Hospital Hemodialysis Center in Izmir. Patients: Forty patients receiving hemodialysis treatment. Interventions: Nine sessions of reflexology massage will be given to reflex points including the solar plexus, brain, pituitary, thyroid, diaphragm, upper lymphs, lung, spinal cord and adrenal glands. Main Outcome Measures: sleep, anxiety, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Conscious and oriented with no communication problem
* Agreeing to participate in the study
* Receiving hemodialysis treatment 3 times a week for 6 months or more
* Patients who have no problem to apply massage; Those who do not have any skin lesions, burns, pathological diseases related to muscles and bones, phlebitis, embolism or bleeding disorder.

Exclusion Criteria:

* Patients who have received hemodialysis treatment for less than 6 months.
* Patients with diabetic neuropathy
* Those who have any skin lesions, burns, open wounds, muscle and bone-related pathological disease, phlebitis, embolism or bleeding disorder in the foot.
* Patients with infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
sleep | nine sessions of foot reflexology massage will be given to reflex points including the solar plexus, brain, pituitary, thyroid, diaphragm, upper lymphs, lung, spinal cord and adrenal glands for 3 weeks.
  improvement in sleep quality. The patients' sleep quality score were collected by the Richard-Campbell Sleep Questionnaire. The scale has a 100-mm line with words describing the poorest possible sleep (0 mm) to the best possible sleep (100 mm).

SECONDARY OUTCOMES:
anxiety | nine sessions of foot reflexology massage will be given to reflex points including the solar plexus, brain, pituitary, thyroid, diaphragm, upper lymphs, lung, spinal cord and adrenal glands for 3 weeks.
  reduce anxiety. The patients' anxiety score data were collected by the State Anxiety Inventory. It is a 20-item scale. The scores in the inventory range from 20 to 80. Higher points show a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Gürol Arslan, PhD, Principal Investigator — Associate professor
Locations (1):
- Başkent University, İzmir Çiğli Dialysis Center, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No